CLINICAL TRIAL: NCT06977659
Title: Early Norepinephrine in Trauma Patients With Hemorrhagic Shock (ENTHeS Trial): A Randomized Open-label Clinical Trial
Brief Title: Early Norepinephrine in Trauma Patients With Hemorrhagic Shock
Acronym: ENTHeS
Status: Enrolling by invitation | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Visarat Palitnonkiat (Other)
Collaborators: Siriraj Hospital (Other)
Responsible Party: Sponsor-Investigator, Visarat Palitnonkiat, Faculty of Medicine Ramathibodi Hospital, Ramathibodi Hospital
Organization: Ramathibodi Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MURA2025/335
Record Dates: First submitted 2025-05-07; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Trauma, Multiple
Keywords: Trauma; Norepinephrine; Blood transfusion
MeSH Terms: conditions — Multiple Trauma; Wounds and Injuries | interventions — Norepinephrine

STUDY DESIGN:
Intervention Model Description: After the trauma team notifies the nurse about the patient's enrollment, an independent nurse opens an opaque sealed envelope (randomization). Afterward, he or she will prepare the drug (norepinephrine or placebo) according to the assigned group and send it to the trauma bay/ ward. Both norepinephrine preparation and matched placebo will be given intravenously at the rate of 10ml/h.
Masking Description: The independent nurse prepares the drug (norepinephrine or placebo) according to the randomization code associated with the study ID and then sends it to the trauma bay. The appearance of both norepinephrine and placebo preparations will be identical. Both patients and physicians will remain blinded after the intervention assignment. An emergency unblinding service is available if the clinician believes that clinical management depends on knowing whether the patient received norepinephrine or placebo. Attending physicians will also be unblinded in the event of serious adverse events that require discontinuation of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Norepinephrine (Active Comparator): Norepinephrine bitartrate (LEVOPHEDR, Pfizer inc.) 4 mg/4ml + 5% Dextrose in water 246 ml (total volume 250 ml, final concentration 16 mcg/ml) infuses intravenously via a central catheter or peripheral line with the rate of 10 ml/h (equivalent to 0.05 mcg/kg/min for a 50-kg patient). The drug will be initiated within 1 hour after randomization, infused for 24 hours after randomization, and then discontinued.
  Interventions: Drug: Norepinephrine
- Placebo (Placebo Comparator): 5% Dextrose in water 250 ml infused intravenously at a rate of 10 ml/h. The drug will be initiated within 1 hour after randomization, infused for 24 hours after randomization, and then discontinued.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Norepinephrine — Norepinephrine bitartrate (LEVOPHEDR, Pfizer inc.) 4 mg/4ml + 5% Dextrose in water 246 ml (total volume 250 ml, final concentration 16 mcg/ml) infuses intravenously via a central catheter or peripheral line with the rate of 10 ml/h (equivalent to 0.05 mcg/kg/min for a 50-kg patient). The drug will be initiated within 1 hour after randomization, infused for 24 hours after randomization, and then discontinued.
  Arms: Norepinephrine
Drug: Placebo — 5% Dextrose in water 250 ml infused intravenously at a rate of 10 ml/h. The drug will be initiated within 1 hour after randomization, infused for 24 hours after randomization, and then discontinued.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if norepinephrine works to treat trauma patients with hemorrhagic shock. It will also learn about the safety of norepinephrine. The main questions it aims to answer are:

Does norepinephrine affect the short-term mortality (24-hour mortality)? Does norepinephrine affect the long-term mortality (30-day mortality), survival with favorable outcome, total volume of blood product and crystalloid given in 24 hours, estimated blood loss within 24 hours, resuscitation-related complications, and length of ICU and hospital stay? What medical problems do participants have when receiving norepinephrine? Researchers will compare norepinephrine to a placebo (a look-alike substance that contains no drug) to see if norepinephrine works to treat trauma patients with hemorrhagic shock.

Participants will:

Receive norepinephrine or a placebo intravenously within 1 hour after randomization, infused for 24 hours after randomization, and then discontinued.

Patients are monitored for outcomes and adverse events.

DETAILED DESCRIPTION:
Study Population: Adult trauma patients with hemorrhagic shock

Inclusion Criteria:

1. Adult trauma patients aged 18 to 65 years
2. Significant bleeding from traumatic events including

   1. Exsanguinous external bleeding (500 ml or more), or
   2. Evidence of internal bleeding (e.g., FAST positive, hemothorax, or bleeding seen on CT scan)
3. Hemorrhagic shock is defined as:

   1. Hypotensive event suspected from hemorrhagic shock, characterized by

      * Systolic blood pressure less than 90 mmHg,
      * Mean arterial pressure less than 65 mmHg, or
      * A decrease in blood pressure from baseline more than 30 mmHg (as recorded in the trauma bay, resuscitation room of the emergency department at Ramathibodi Hospital, trauma unit at Siriraj Hospital, or trauma ward/ ICU) OR
   2. Signs of shock, including:

      * Capillary refill time greater than 2 seconds,
      * Base excess less than -6 mEq/L,
      * Lactate level greater than 2 mmol/L)

Exclusion criteria

1. Prehospital cardiopulmonary resuscitation or cardiopulmonary resuscitation at the trauma bay.
2. Persistent shock for more than 12 hours prior to randomization.
3. Severe traumatic brain injury with Glasgow Coma Scale (GCS) score less than 9 (GCS 3-8)
4. Traumatic limb injury with acute limb ischemia
5. A history of limb ischemia, chronic heart disease, chronic lung disease, or chronic renal disease
6. Pregnant patients
7. Documented "Do Not Resuscitate" (DNR) order or who declined life-sustaining intervention before randomization
8. Allergic to norepinephrine or contraindications for its use (e.g., peripheral vascular thrombosis, mesenteric thrombosis, and fatal tachyarrhythmia)
9. Current use of ergotamine, monoamine oxidase inhibitors (MAOIs), or tricyclic antidepressants (TCAs)
10. Prior vasopressor administration before randomization.
11. Weight less than 30 kilograms (Extremely low body weight may increase the risk of weight-based dosing issues)

The independent nurse prepares the drug (norepinephrine or placebo) according to the randomization code associated with the study ID and then sends it to the trauma bay. The appearance of both norepinephrine and placebo preparations will be identical. Both patients and physicians will remain blinded after the intervention assignment. An emergency unblinding service is available if the clinician believes that clinical management depends on knowing whether the patient received norepinephrine or placebo. Attending physicians will also be unblinded in the event of serious adverse events that require discontinuation of the study.

Intervention group:

* Drug: Norepinephrine bitartrate (LEVOPHEDR, Pfizer inc.) 4 mg/4ml + 5% Dextrose in water 246 ml (total volume 250 ml, final concentration 16 mcg/ml) infuses intravenously via a central catheter or peripheral line with the rate of 10 ml/h (equivalent to 0.05 mcg/kg/min for a 50-kg patient). The drug will be initiated within 1 hour after randomization, infused for 24 hours after randomization, and then discontinued.
* If at any time during the infusion the patient's systolic blood pressure is above 160 mmHg30 for 10 min, the infusion will be held up for 30 min. After 30 min, if the SBP is less than 160, the infusion was resumed at a rate of 5ml/h (50%). If the SBP remains less than 160, the infusion will be increased to the original dose of 10ml/h (100%).
* Medical device: The norepinephrine preparation or placebo will be infused with each institute's syringe or infusion pump available. The ENTHES solution will be infused through a separate peripheral IV access.

Control group:

Placebo: 5% Dextrose in water 250 ml infused intravenously with a rate of 10 ml/h

Both groups will receive standard trauma care based on ATLS guidelines, which includes the following: 2 large-bore intravenous access, a bolus of warm isotonic crystalloids (500-1,000 mL), and consideration of tranexamic acid based on the duration of injury. Bleeding will be controlled, and laboratory investigations, such as iStat, arterial blood gas, base excess, complete blood count, coagulogram, will be performed. The massive transfusion protocol may also be considered. If the attending physician wishes to add or increase the vasopressor dose, it will be prepared separately.

After the ENTHES solution has been infused for 24 hours, if the patients experiences hypotension, either noninvasive or invasive monitoring will be used to assess fluid responsiveness, and standard management will be provided based on the attending physician's judgement. If the cause of hypotension is due to decreased vascular resistance, a vasoactive agent such as norepinephrine or epinephrine will be initiated.

Primary outcome: 24-hour mortality

Secondary outcome: 30-day mortality, survival with favorable outcome at 30 days (defined as modified Rankin Score (mRS) of 0-3), survival to hospital discharge, death in OR, the cumulative volume of blood product in milliliter (ml) transfused within 24 hours (included PRBC, FFP, platelets, and cryoprecipitates), the total volume of crystalloid (in mL) infused within 24 hours, total urine output within 24 hours, vital signs trending over 24 hours, Intake/ output balance over 24 hours, tissue perfusion parameters (e.g., serum lactate in mmol/L, base deficit in mEq/L), estimated blood loss in ml within 24 hours, length of ICU stays (in days), length of hospital stays (in days), and length of mechanical ventilation.

Safety outcome: Adverse events of norepinephrine (e.g. arrhythmia, hypertensive emergency, acute mesenteric ischemia, peripheral vascular ischemia, and drug allergy) and other adverse events (ARDS (according to a new global definition of ARDS 2023), transfusion complication, AKI (KDIGO 2012), acute myocardial infarction, surgical site or wound infection, ventilator-associated pneumonia, compartment syndrome, deep vein thrombosis, pulmonary embolism, rhabdomyolysis and gastrointestinal bleeding)

Discontinuation/withdrawal criteria:

1. The participant or his relative's withdrawal requests
2. The attending physician's judgement to withdraw from the study

ELIGIBILITY:
Inclusion Criteria:

1. Adult trauma patients aged 18 to 65 years
2. Significant bleeding from traumatic events including

   1. Exsanguinous external bleeding (500 ml or more), or
   2. Evidence of internal bleeding (e.g., FAST positive, hemothorax, or bleeding seen on CT scan)
3. Hemorrhagic shock is defined as:

   1. Hypotensive event suspected from hemorrhagic shock, characterized by

      * Systolic blood pressure less than 90 mmHg,
      * Mean arterial pressure less than 65 mmHg, or
      * A decrease in blood pressure from baseline more than 30 mmHg (as recorded in the trauma bay, resuscitation room of the emergency department at Ramathibodi Hospital, trauma unit at Siriraj Hospital, or trauma ward/ ICU) OR
   2. Signs of shock, including:

      * Capillary refill time greater than 2 seconds,
      * Base excess less than -6 mEq/L,
      * Lactate level greater than 2 mmol/L)

Exclusion Criteria:

1. Prehospital cardiopulmonary resuscitation or cardiopulmonary resuscitation at the trauma bay.
2. Persistent shock for more than 12 hours prior to randomization.
3. Severe traumatic brain injury with Glasgow Coma Scale (GCS) score less than 9 (GCS 3-8)
4. Traumatic limb injury with acute limb ischemia
5. A history of limb ischemia, chronic heart disease, chronic lung disease, or chronic renal disease
6. Pregnant patients
7. Documented "Do Not Resuscitate" (DNR) order or who declined life-sustaining intervention before randomization
8. Allergic to norepinephrine or contraindications for its use (e.g., peripheral vascular thrombosis, mesenteric thrombosis, and fatal tachyarrhythmia)
9. Current use of ergotamine, monoamine oxidase inhibitors (MAOIs), or tricyclic antidepressants (TCAs)
10. Prior vasopressor administration before randomization.
11. Weight less than 30 kilograms (Extremely low body weight may increases the risk of weight-based dosing issues)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-07-17 (Estimated); Study Completion 2027-08-18 (Estimated)

PRIMARY OUTCOMES:
24-hour mortality | From enrollment to the end of treatment at 24 hour
  The outcome will be analyzed 24 hours after the patient is enrolled.

SECONDARY OUTCOMES:
30-day mortality | From enrollment to 30 days after treatment.
  The outcome will be analyzed at 30 days after the patient is enrolled.
Survival with favorable outcome at 30 days | From enrollment to 30 day after treatment.
  The favorable outcome is defined as a modified Rankin Score (mRS) of 0-3. A modified Rankin Scale (mRS) ranges from 0 to 6, with lower scores indicating better outcomes.
The cumulative volume of blood product within 24 hours | From enrollment to the end of treatment at 24 hour.
  Blood volume is reported in milliliter (mL) included RBCs, FFP, platelet, and cryoprecipitate)

CONTACTS AND LOCATIONS:
Locations (2):
- Thailand (2):
  - Faculty of Medicine Ramathibodi Hospital, Bangkok
  - Faculty of Medicine Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) that could identify patients will not be shared. Only de-identified supporting data relevant to the study will be made available to collaborating centers upon reasonable request, for the purposes of academic research and secondary analyses related to the original study objectives. Data will be shared via secure, institutional data-sharing mechanisms. All requests will be reviewed by the principal investigator and the study's data access committee based on scientific merit, ethical considerations, and alignment with the original study scope. Shared data will be deleted by the recipient institutions within five years after publication of the study findings

REFERENCES:
- [Background] Harrois A, Baudry N, Huet O, Kato H, Dupic L, Lohez M, Ziol M, Vicaut E, Duranteau J. Norepinephrine Decreases Fluid Requirements and Blood Loss While Preserving Intestinal Villi Microcirculation during Fluid Resuscitation of Uncontrolled Hemorrhagic Shock in Mice. Anesthesiology. 2015 May;122(5):1093-102. doi: 10.1097/ALN.0000000000000639. PMID 25782753
- [Background] Cohn SM, DeRosa M, McCarthy J, Song J, White C, Louden C, Ehler B, Michalek J, Landry DW. Characterizing vasopressin and other vasoactive mediators released during resuscitation of trauma patients. J Trauma Acute Care Surg. 2013 Oct;75(4):620-8. doi: 10.1097/TA.0b013e31829eff31. PMID 24064875
- [Background] Cohn SM, McCarthy J, Stewart RM, Jonas RB, Dent DL, Michalek JE. Impact of low-dose vasopressin on trauma outcome: prospective randomized study. World J Surg. 2011 Feb;35(2):430-9. doi: 10.1007/s00268-010-0875-8. PMID 21161222